CLINICAL TRIAL: NCT01194466
Title: The Influence of TENS on Mucositis Pain and Function in Head and Neck Cancer Patients: A Randomized and Placebo-Controlled Double Blind Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) and Head and Neck Cancer Pain (HNC) (TENS & HNC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer E. Lee (Other)
Responsible Party: Sponsor-Investigator, Jennifer E. Lee, Post Doctoral Research Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: University of Iowa 201009732
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Head Cancer; Neck Cancer; Pain
Keywords: Head and Neck Cancer; Oral Cancer; Laryngeal Cancer; Oropharyngeal Cancer; Transcutaneous Electrical Nerve Stimulation (TENS); Oral Mucositis; Pain; Function; TENS; Functional Pain; Non-pharamcologic; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Mouth Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms; Stomatitis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active TENS (Active Comparator): Active high frequency TENS will be use for Active TENS.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Placebo (low intensity) TENS (Experimental): Placebo TENS will be applied for one arm of the study
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- No Treatment (Sham Comparator): TENS unit in place but not turned on
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Four adhesive electrodes (1.375in x 1.375in) will be placed bilaterally on the: 1) temporomandibular joint (1/3rd of distance between ear and nose); and 2) upper neck area (2cm from spine, i.e., Cervical 1 and 2).
  Other Names: EMPI Select

SUMMARY:
The overall goal of this study is to examine the effect of a single dose of TENS on mucositis pain and function secondary to head and neck radiation therapies. Oral mucositis is an extremely debilitating, unpreventable condition (inflammation, ulcers, bleeding in the mouth, nose, and throat) that causes significant pain, functional impairment, and diminished quality of life. Head and neck cancers pose specific challenges to effective pain management and past studies suggest the use of effective non-pharmacologic strategies such as TENS may be particularly beneficial for avoiding sources of acute and chronic pain, thereby improving quality of life. The investigators hypothesize that a single dose of TENS will decrease pain and improve function and quality of life in head and neck cancer patients. This project is particularly innovative because it is the first known study to examine the efficacy of TENS, an established safe, inexpensive and easy-to-use non-pharmacologic pain management intervention, for treating acute oral mucositis pain. The investigators research translates bench (animal model) science to human subjects using an interdisciplinary approach to pain management. Establishing whether TENS is effective for reducing mucositis pain is a critical first step toward establishing an effective, non-pharmacologic pain relief intervention for mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck Cancer Diagnosis
* Oral mucositis diagnosis

Exclusion Criteria:

* TENS use ≤ 5 years
* Pacemaker
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05-15 (Actual); Primary Completion 2012-08-14 (Actual); Study Completion 2012-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Lee, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized, double-blinded, and placebo controlled study was conducted between May 2011 and August 2012 at the University of Iowa Hospitals and Clinics (Clinical-Trials.gov identifier, NCT01194466)
Pre-assignment Details: Study exclusion criteria were (1) TENS use within 5 years, (2) conditions precluding TENS use (pacemaker, nickel allergy), (3) pain intensity less than 1 of 10 with rest or swallowing, (4) sensory impairment (could not identify sharp and dull stimuli on face), and/or (5) inability to read, write, or follow directions.
Groups:
- Order: Active, Placebo, No TENS: Active high frequency TENS will be used visit 1 Washout 6 days Placebo for visit 2- 7 days after visit 1 Washout for 6 days No tens visit 3- 7 days after visit 2
- Order: Placebo, Active, No TENS: Placebo low frequency TENS will be used visit 1 Washout 6 days Active high intensity TENS for visit 2- 7 days after visit 1 Washout for 6 days No tens visit 3- 7 days after visit 2
- Order: No TENS, Active, Placebo: No TENS will be used visit 1 Washout 6 days Active high intensity TENS for visit 2- 7 days after visit 1 Washout for 6 days Placebo Low Intensity TENS visit 3- 7 days after visit 2
Period: Overall Study
Arm/Group | Order: Active, Placebo, No TENS | Order: Placebo, Active, No TENS | Order: No TENS, Active, Placebo
Started | 14 | 14 | 13
Completed | 14 | 14 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants' characteristics, prior to first treatment
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity in Head/Neck Cancer Area: 10cm Visual Analog Scale (VAS)
Description: Participants rated 0-10 pain intensity in head/neck cancer area using one number (where their disease was located) by a vertical line on a horizontal 10-cm visual analog scale (VAS) from 0 "no pain" to 10 "worst possible pain." Possible scores ranged from 0-10 (10=worse pain). VAS was assessed two times each visit: (1) Pre-VAS: start of visit, (2) Post-VAS: end of the visit. The outcome measure was each person's change in pain: Pre-VAS minus Post-VAS, to create VAS change score. An average of all participants' VAS change score was calculated for each TENS condition (Active, Placebo, No TENS) and used as the dependent measure.
Time Frame: The change in VAS pain score was assessed within one study visit for each of the 3 study TENS conditions
Population: The sample was adults (18 or greater) years old with oropharyngeal or laryngeal cancer.
Measure: Mean (Standard Deviation); unit: change units on a VAS scale
Groups:
- Active TENS: Each participant received an Active TENS intervention at one clinic visit, separated approximately one week from the other 2 TENS condition visits. In other words, all participants received the Active TENS condition. Active TENS was delivered for 30 minutes at a frequency of 125Hz and a pulse duration of 100 2s on continuous mode output (calibrated using an oscilloscope before the study). Transcutaneous electrical nerve stimulation intensity was increased by the allocator until patients reported a ''maximally strong but comfortable sensation'' to ensure an analgesic effect.
- Placebo TENS: Each participant received an Placebo TENS intervention at one clinic visit, separated approximately one week from the other 2 TENS condition visits. In other words, all participants received the Placebo TENS condition. Placebo TENS parameters were identical to active TENS (125 Hz, 100 2s). A novel, transient placebo TENS unit, previously tested and validated, was used. The intensity was increased until patients first felt ''any sensation at all (sensory threshold)'' in any electrode (ie, they did not have to reach sensory threshold in all electrodes). The placebo device then provided a current for 30 seconds and decreased gradually over 15 seconds to 0 output (ie, 45 seconds from the first sensory threshold). An indicator light remained on for the remainder of the visit so it appeared to the participant and outcomes assessor that the unit was still producing current.
- No TENS: Each participant received a No TENS intervention at one clinic visit, separated approximately one week from the other 2 TENS condition visits. In other words, all participants received the No TENS condition. No TENS parameters were identical to active and placebo TENS, except that (1) the unit was never turned on and (2) participants were told that the unit was not on.
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 40 | 40 | 40
change units on a VAS scale | -1.4 (1.3) | -0.6 (1.1) | 0.1 (0.9)

ADVERSE EVENTS:
Groups:
- Low Intensity TENS: Low Intensity TENS will be applied for one arm of the study
  Transcutaneous Electrical Nerve Stimulation (TENS): Four adhesive electrodes (1.375in x 1.375in) will be placed bilaterally on the: 1) temporomandibular joint (1/3rd of distance between ear and nose); and 2) upper neck area (2cm from spine, i.e., Cervical 1 and 2).
Arm/Group | Active TENS | Low Intensity TENS | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No